CLINICAL TRIAL: NCT03211754
Title: Changes on Anthropometric Measures and Anti-inflammatory Markers by a PUFAs Enriched Diet in Obese Subjects
Brief Title: Anthropometric Measures and Anti-inflammatory Markers by a PUFAs Enriched Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Elva Perez-Luque, Profesor-Investigator, Universidad de Guanajuato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UGuanajuato
Record Dates: First submitted 2017-06-30; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: Walnuts; almonds; adiponectin; lipocalin-2; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obese patients (Experimental): Treatment for 8 weeks
  Interventions: Dietary Supplement: walnuts and almonds

INTERVENTIONS:
Dietary Supplement: walnuts and almonds — The subjects consumed 15g of walnuts and 15g of almonds/day for 8 weeks

SUMMARY:
In this work, the investigators report the effects of consume of 15g walnuts and 15g almonds for 8 week on weight, waist and hip circumferences, body mass index, fat mass, serum LDL-cholesterol adiponectin, lipocalin-2 concentration and fatty acids profile.

DETAILED DESCRIPTION:
The study consists of a diet-intervention in a single group under-free-living conditions. The diet was enriched with 15g of almonds and 15g of walnuts per day for eight weeks, supplied directly to the patient by the researcher. This amounts of walnuts and almonds contain polyunsaturated fatty acids of approximately 2.02g of omega 3 (alpha-linolenic acid) and 11.1g of omega 6 (linoleic acid) mostly. In a period of 14 months, the investigators recruited forty-eight sedentary subjects of 30 to 50 years old, and body mass index between 30 and 34.9 kg/m2, without evidence of chronic degenerative, infectious or neoplastic diseases, neither medication nor actually dietary treatment, and a physical level of exercise < 2 hours/week. All participants gave their written informed consent to participate in the study. The study was approved by the Institutional Ethics Committee of the Universidad de Guanajuato.

Collected data included the clinical-nutritional history, 24-hour recalls, and the International Physical Activity Questionnaire was applied to evaluate if subjects were sedentary. The dietary intake evaluation was estimated in kilocalories/day, the amount and type of macronutrients according to the database of United States Department of Agriculture and the National Institute of Public Health (Mexico). In order to evaluate adherence to the diet, volunteers were visited every two weeks to carry out three 24-hour recalls (two on weekdays and one on weekends). Positive Adherence to the diet plan was considered when the food consumption, walnuts and almonds were not modified more than ± 20% of the amount indicated by the researcher.

The investigators recorded the anthropometric measures, body composition, and measured serum glucose, lipid profile, insulin, lipocalin 2, high sensitivity C-reactive protein, adiponectin, and fatty acids profile, which were analyzed at the baseline and after dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

- obesity grade I

Exclusion Criteria:

* Subjects did not have evidence of chronic degenerative, infectious or neoplastic disease.
* Lack of adherence to the diet and consumption of walnuts and almonds

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Metabolics Changes | 8 weeks
  fatty acids in percentage

SECONDARY OUTCOMES:
Significant decreases on all adiposity measures | 8 weeks
  Weight in kilograms
Significant decreases on all adiposity measures | 8 weeks
  height in meters
Significant decreases on all adiposity measures | 8 weeks
  waist circumference in centimeters
Significant decreases on all adiposity measures | 8 weeks
  hip circumference in centimeters
Significant decreases on all adiposity measures | 8 weeks
  fat mass in percentage
Significant decreases on all adiposity measures | 8 weeks
  Weight and height will be combined to report BMI in kg/m2
Metabolics Changes | 8 weeks
  Glucose in mg/dL
Metabolics Changes | 8 weeks
  total Cholesterol in mg/dL
Metabolics Changes | 8 weeks
  LDL-cholesterol in mg/dL
Metabolics Changes | 8 weeks
  HDL-cholesterol in mg/dL
Metabolics Changes | 8 weeks
  triglycerides in mg/dL
Metabolics Changes | 8 weeks
  Lipocalin-2 in mg/mL
Metabolics Changes | 8 weeks
  Insulin in pmol/L
Metabolics Changes | 8 weeks
  High sensitivity C-reactive protein in mg/L
Metabolics Changes | 8 weeks
  adiponectin in microg/mL